CLINICAL TRIAL: NCT06813716
Title: Comparison of the Acute Effects of Two Neoprene Knee Sleeves on Balance and Pain in Knee Osteoarthritis: A Randomized, Single-Blinded, Prospective Study
Brief Title: Acute Effects of Two Neoprene Knee Sleeves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Fulya Bakılan, Associate Professor, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ESOGUFtr1
Record Dates: First submitted 2025-01-31; First posted 2025-02-07 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthristis
Keywords: Balance, knee sleeve, osteoarthritis, posturography
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 : consisted of 30 patients wearing elastic neoprene knee sleeve (Active Comparator)
  Interventions: Other: Neoprene elastic knee sleeve
- group 2 consisted of 30 patients wearing neoprene knee sleeve with four metal supports (Active Comparator)
  Interventions: Other: Neoprene elastic knee sleeve with metal supports

INTERVENTIONS:
Other: Neoprene elastic knee sleeve — We hypothesized that a neoprene elastic knee sleeve with metal supports would have a greater acute effect on balance and pain than a neoprene elastic sleeve. The first study to evaluate the acute effects of 2 different knee sleeves on pain and balance.
  Arms: Group 1 : consisted of 30 patients wearing elastic neoprene knee sleeve
Other: Neoprene elastic knee sleeve with metal supports — We hypothesized that a neoprene elastic knee sleeve with metal supports would have a greater acute effect on balance and pain than a neoprene elastic sleeve. The first study to evaluate the acute effects of 2 different knee sleeves on pain and balance.
  Arms: group 2 consisted of 30 patients wearing neoprene knee sleeve with four metal supports

SUMMARY:
This study aimed to evaluate the immediate effects of two different types of elastic neoprene knee sleeves on balance and pain in patients with knee osteoarthritis (KOA). One knee sleeve was a standard elastic neoprene sleeve, while the other had four metal supports for additional stability.

In this randomized controlled study, 60 patients (50 females, 10 males) diagnosed with KOA were divided into two groups:

Group 1: Wore a standard elastic neoprene knee sleeve Group 2: Wore a neoprene knee sleeve with four metal supports

Each participant underwent clinical assessments before and after wearing the knee sleeve. The following tests were used:

Balance Assessments:

Berg Balance Scale (BBS): Measures overall balance ability. Timed Up and Go (TUG) Test: Evaluates mobility and fall risk. Functional Reach Test (FRT): Assesses stability by measuring how far a person can reach forward.

Fall Index (Tetrax® posturography): Provides an objective measure of fall risk.

Pain Assessment:

Visual Analog Scale (VAS): Measures the intensity of pain.

Further long-term studies are necessary to determine whether these immediate benefits persist over time.

DETAILED DESCRIPTION:
KOA is a common joint disorder that leads to pain, stiffness, and impaired balance, increasing the risk of falls. Knee sleeves are often used as supportive devices to provide stability and reduce pain. However, there is limited evidence on their effectiveness in improving balance and reducing pain in KOA patients.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic knee osteoarthritis grade 2 (mild) or 3 (moderate) according to Kellgren-Lawrence scale,
* Knee muscle strength of 4 and above and those who voluntarily participated in the study
* Signed the informed consent form

Exclusion Criteria:

* Patients with arthroscopy of the knee joint within the last 1 year, knee and/or hip replacement,
* Limitation of joint range of motion,
* History of inflammatory rheumatic disease,
* History of vestibular and cerebellar disease,
* Visual loss of less than 2/10 in both eyes,
* History of diseases of the central and peripheral nervous system (Parkinson's disease, stroke, ataxia, dementia, multiple sclerosis, peripheral neuropath etc.)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
The Berg Balance Scale (BBS) | Assessments were performed before and immediately after wearing the knee sleeves
  Total score is between 0-56. 56 points indicates perfect balance

SECONDARY OUTCOMES:
Timed Up and Go (TUG) | Assessments were performed before and immediately after wearing the knee sleeves
  This test, which evaluates balance function is reported that a threshold value above 14 seconds predicts falls with high sensitivity and specificity.
Functional Reach Test (FRT) | Assessments were performed before and immediately after wearing the knee sleeves
  15 cm or less indicates a significantly increased risk of falling, while 15 to 25 cm indicates a moderate risk of falling.
Fall Index, calculated using posturography (Tetrax®) | Assessments were performed before and immediately after wearing the knee sleeves
  100 indicates the lowest risk of falling, while 0 indicates the highest risk of falling.
the Visual Analog Scale (VAS) | Assessments were performed before and immediately after wearing the knee sleeves
  Patients were required to indicate the level of pain they were experiencing on a scale of 0 to 10, with 0 representing no pain and 10 representing the most intense pain they had ever felt.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskişehir Osmangazi University Department of Physical Medicine and Rehabilitation, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided